CLINICAL TRIAL: NCT05693051
Title: Use of Prone Position Ventilation (PPV) in Danish Patients With COVID-19 Induced Severe Adult Respiratory Distress Syndrome (ARDS) Treated With Veno-Venous Extracorporeal Membrane Oxygenation (VV-ECMO)
Brief Title: Use of Prone Position Ventilation in Danish Patients With COVID-19 Induced Severe ARDS Treated With VV-ECMO
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Lind Jørgensen, Consultant, PhD, principal investigator, Rigshospitalet, Denmark
Other Study IDs: 20049299-PPV
Record Dates: First submitted 2023-01-18; First posted 2023-01-20 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: ARDS, Human; Extracorporeal Membrane Oxygenation; COVID-19 Acute Respiratory Distress Syndrome; Prone Position; Adverse Event
Keywords: ARDS; VV-ECMO; Prone position ventilation; Adverse Events
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prone position ventilation — Turning the patient prone for 16 hours

SUMMARY:
Prone position ventilation was used 220 times in 44 out of 68 patients with severe COVID-19 induced ARDS treated with VV-ECMO. PPV treated patients did not benefit from PPV and the incidence of PPV related adverse events was high

DETAILED DESCRIPTION:
Purpose: To describe the use and effects of prone position ventilation (PPV) in patients with COVID-19 induced Adult Respiratory Distress Syndrome (ARDS), treated with Veno-Venous Extracorporeal membrane oxygenation (VV-ECMO).

Methods: Nationwide retrospective analysis of all COVID-19 patients in Denmark from March 2020 - December 2021with severe ARDS and need of VV-ECMO treatment. Data on the number of patients treated with PPV, number of PPV-events, timing, the time spent in prone position, physiological response types, adverse events and outcomes are reported.

ELIGIBILITY:
Inclusion Criteria: patients with COVID-19 induced severe ARDS accepted for and treated with VV-ECMO in Denmark

-

Exclusion Criteria:

* none

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a nationwide retrospective cohort study of a cohort of 68 patients with PCR confirmed SARS-Cov-2 ARDS, treated with V-V ECMO in the two VV-ECMO centers in Denmark: Aarhus University Hospital in west Denmark and University Hospital Rigshospitalet in Copenhagen, East Denmark. Patients were admitted in the period from 17. March 2020 to 31. December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
90 day mortality | 90 days
  all cause mortality 90 days after ECMO start

SECONDARY OUTCOMES:
Time-to-wean | From start of ECMO treatment to succesful weaning from ECMO
  Time from ECMO start to succesful weaning from ECMO
Recruitment Response to prone position ventilation | from prone position start to prone position end
  lung recruitment
Oxygenation Response to prone position ventilation | from prone position start to prone position end
  Oxygenation

OTHER OUTCOMES:
Adverse Events | From ECMO start to ECMO end (all causes)
  Number and nature of adverse events related to prone position ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke L Jorgensen, M.D, Principal Investigator — Department of CardioThoracic Anesthesia and Intensive Care, Rigshospitalet University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, CardioThoracic Intensive care Unit, Aarhus
  - University Hospital Rigshospitalet, department of CardioThoracic Anaesthesia and Intensive Care, Copenhagen

IPD SHARING:
Plan to Share IPD: No